CLINICAL TRIAL: NCT06897475
Title: A Parallel-Group Treatment, Phase 2, Double-Blind Study of Once-Weekly Subcutaneous LY3457263 Compared to Placebo in Participants With Type 2 Diabetes Mellitus on a Stable Dose of Semaglutide or Tirzepatide Who Failed to Achieve HbA1c Goal
Brief Title: A Study of LY3457263 Compared With Placebo in Participants With Type 2 Diabetes on a Stable Dose of Semaglutide or Tirzepatide
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27344; 2024-520328-27-00 (EU CTIS Number); J1R-MC-GZFD (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-03-25; First posted 2025-03-27 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Type 2 Diabetes
Keywords: Obesity; Overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3457263 Dose 1 (Experimental): Participants will receive LY3457263 subcutaneously (SC)
  Interventions: Drug: LY3457263
- LY3457263 Dose 2 (Experimental): Participants will receive LY3457263 SC
  Interventions: Drug: LY3457263
- LY3457263 Dose 3 (Experimental): Participants will receive LY3457263 SC
  Interventions: Drug: LY3457263
- Placebo (Placebo Comparator): Participants will receive placebo SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3457263 — Administered SC
  Arms: LY3457263 Dose 1; LY3457263 Dose 2; LY3457263 Dose 3
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure the change in hemoglobin A1c (HbA1c) with LY3457263 compared with placebo in participants with type 2 diabetes who are not at HbA1c goal when treated with a stable dose of semaglutide or tirzepatide. Participation in the study will last about 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes
* Have HbA1c ≥7.5% to ≤10.5% at screening
* Have a body mass index (BMI) of ≥27 kilograms per square meter (kg/m2) at screening
* Have had a stable body weight for the three months prior to screening
* On stable treatment dose of one of the following incretins for at least three months prior to screening:

  * Injectable semaglutide (1 and 2 milligram (mg))
  * Injectable tirzepatide (5, 7.5, 10, 12.5 and 15 mg)

Exclusion Criteria:

* Have type 1 diabetes, latent autoimmune diabetes, or history of ketoacidosis or hyperosmolar coma
* Have a prior or planned surgical treatment for obesity
* Have any of the following cardiovascular conditions within three months prior to screening:

  * acute myocardial infarction
  * cerebrovascular accident (stroke)
  * unstable angina, or
  * hospitalization due to congestive heart failure
* Have used insulin to control blood glucose within the past year (short-term use allowed)
* Current use of prohibited oral antihyperglycemic medication (OAM) (including but not limited to, Dipeptidyl Peptidase IV Inhibitors (DPP-4i) and meglitinides) may be randomized if the prohibited OAM treatment was discontinued at least 3 months prior to screening

  * If participant has been on stable doses (for at least three months) of up to three permitted OAMs (limited to metformin, sodium-glucose cotransporter-2 (SGLT2) inhibitors, alpha-glucosidase inhibitors, sulfonylurea, and/or thiazolidinediones (TZD), they are permitted to participate in the study
* Have taken any medications or alternative remedies for weight loss within three months prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 24

SECONDARY OUTCOMES:
Change from Baseline in Fasting Serum Glucose | Baseline, Week 24
Percent Change from Baseline in Body Weight | Baseline, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (56):
- United States (20):
  - Helios Clinical Research - Phoenix, Phoenix, Arizona
  - Wolverine Clinical Trials, Santa Ana, California
  - Renstar Medical Research, Ocala, Florida
  - Oviedo Medical Research, Oviedo, Florida
  - Balanced Life Health Care Solutions/SKYCRNG, Lawrenceville, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Elite Clinical Trials, Rexburg, Idaho
  - Investigators Research Group, Brownsburg, Indiana
  - Richmond University Medical Center, Staten Island, New York
  - Southgate Medical Group, West Seneca, New York
  - Lucas Research, Inc., Morehead City, North Carolina
  - Shelby Clinical Research, Shelby, North Carolina
  - Providence Health Partners-Center for Clinical Research, Dayton, Ohio
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - Juno Research, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Texas Diabetes & Endocrinology, P.A., Round Rock, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Eastside Research Associates, Redmond, Washington
- Canada (10):
  - Centricity Research Brampton Endocrinology, Brampton
  - Ecogene-21, Chicoutimi
  - Viacar Recherche Clinique, Greenfield Park
  - Winterberry Research Inc., Hamilton
  - G A Research Associates, Moncton
  - Private Practice - Dr. James Cha, Oshawa
  - Bluewater Clinical Research Group Inc., Sarnia
  - Maple Leaf Research, Toronto
  - Diabetes Heart Research Centre, Toronto
  - Fadia El Boreky Medicine, Waterloo
- Germany (5):
  - InnoDiab Forschung Gmbh, Essen
  - Velocity Clinical Research, Leipzig, Leipzig
  - Gemeinschaftspraxis Dr. Taeschner/Dr. Bonigut, Leipzig
  - Institut für Diabetesforschung GmbH Münster, Münster
  - RED-Institut GmbH, Oldenburg
- Poland (9):
  - Legeartis - Poradnie Specjalistyczne, Bialystok
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk
  - Medyczne Centrum Diabetologiczno Endokrynologiczno Metaboliczne DIAB-ENDO-MET, Krakow
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz
  - Ekamed, Lublin
  - Private Practice - Dr. Robert Witek, Tarnów
  - NBR Polska, Warsaw
  - Szpital Czerniakowski, Warsaw
  - 4 Wojskowy Szpital Kliniczny z Polikliniką SPZOZ, Wroclaw
- Puerto Rico (2):
  - Centro de Endocrinologia Alcantara Gonzalez, Bayamón
  - Mgcendo Llc, San Juan
- United Kingdom (10):
  - FutureMeds - Birmingham, Birmingham
  - Layton Medical Centre, Blackpool
  - Southmead Hospital, Bristol
  - FutureMeds - Liverpool, Bromborough
  - Futuremeds-Newcastle, Newcastle
  - Newquay Health Centre, Newquay
  - George Eliot Hospital, Nuneaton
  - The Adam Practice, Poole
  - Clifton Medical Centre, Rotherham
  - Rame Group Practice, Torpoint

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of LY3457263 Compared with Placebo in Participants with Type 2 Diabetes on a Stable Dose of Semaglutide or Tirzepatide — https://trials.lilly.com/en-US/trial/587456